CLINICAL TRIAL: NCT00958295
Title: Epidemiology of Acute Bacterial Uncomplicated Cystitis in General Practice: Description and Prediction by Urine Dipstick Test
Brief Title: Epidemiology of Acute Bacterial Uncomplicated Cystitis in General Practice
Acronym: BaCyst
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/119/HP
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2012-12

CONDITIONS: Acute Uncomplicated Bacterial Cystitis
Keywords: urinary tract infection; cystitis
MeSH Terms: conditions — Urinary Tract Infections; Cystitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacterial strains isolated in urine cultures
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute uncomplicated bacterial cystitis is common in general practice. Cystitis is at the second raw of antibiotic treatment indications. It has been now recommended not to perform any urine culture for more than 20 years; hence, the bacterial epidemiology of acute uncomplicated cystitis is surprisingly relatively unknown. The available bacteriological data mainly describe the epidemiology of complicated urinary tract infections or upper urinary tract infections, but the causative bacteria and the resistance rates might differ from those of uncomplicated cystitis. As an example, it is unknown to what extent Staphylococcus saprophyticus is the causative agent of uncomplicated cystitis.

Moreover, the urine dipstick test have been evaluated in laboratories. But their interpretation in current practice might not be so easy: in particular, the nitrite detection depends on the bacterial concentration. The nitrite detection, produced in enterobacteriaceae related infections might have therapeutical consequences: trométamol-fosfomycine is almost constantly active on enterobacteriaceae, but ineffective on staphylococci. Knowing the increasing prevalence of fluoroquinolone-resistant enterobacteriaceae, the use of fosfomycin in nitrite positive uncomplicated cystitis might preserve the susceptibility of fluoroquinolones during pyelonephritis.

This study will describe:

* the bacterial epidemiology of acute uncomplicated cystitis in general practice,
* the correlation in between urine dipstick and urine culture in general practice,
* the prediction of enterobacterial infection by the nitrite detection, AND
* the antibiotics prescribed by the practitioners for uncomplicated acute cystitis.

ELIGIBILITY:
Inclusion Criteria:

* female
* >18 years old
* urinary symptoms

Exclusion Criteria:

* fever
* lumbar pain
* co-morbidities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female, no comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2009-03; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Bacterial epidemiology of acute uncomplicated cystitis | march 2010

SECONDARY OUTCOMES:
Comparison of urine dipstick tests and urine culture results | march 2010

CONTACTS AND LOCATIONS:
Overall Officials: Manuel ETIENNE, MD, Principal Investigator — Infectious diseases department, rouen university hospital
Locations (1):
- JULIENNE Pascal, Louviers, France

REFERENCES:
- [Derived] Etienne M, Lefebvre E, Frebourg N, Hamel H, Pestel-Caron M, Caron F; Bacyst Study Group. Antibiotic treatment of acute uncomplicated cystitis based on rapid urine test and local epidemiology: lessons from a primary care series. BMC Infect Dis. 2014 Mar 11;14:137. doi: 10.1186/1471-2334-14-137. PMID 24612927